CLINICAL TRIAL: NCT06097364
Title: A Phase 3, Open-Label, Randomized Study to Compare the Efficacy and Safety of Odronextamab (REGN1979), an Anti-CD20x Anti-CD3 Bispecific Antibody, Combined With Chemotherapy Versus Rituximab Combined With Chemotherapy in Previously Untreated Participants With Follicular Lymphoma (OLYMPIA-2)
Brief Title: A Trial to Learn if Odronextamab Combined With Chemotherapy is Safe and Well-Tolerated and How Well it Works Compared to Rituximab Combined With Chemotherapy for Adult Participants With Follicular Lymphoma
Acronym: OLYMPIA-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-ONC-2075; 2022-502113-28-00 (Other: EUCT Number)
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Follicular Lymphoma (FL)
Keywords: Non-Hodgkin lymphomas (NHL); Relapsed or Refractory (R/R) FL; B-cells NHL (B-NHL); Untreated FL; Odronextamab
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Odronextamab + Chemotherapy (Experimental): Part 1 of the study includes ordonextamab dose escalation for participants with previously untreated FL and relapsed/refractory FL (Part 1A only) followed by a randomized exploration of 2 regimens of odronextamab (Odro) and cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP) with the objective of dose optimization (Part 1B) in previously untreated patients with FL.
  Interventions: Drug: Odronextamab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone/Prenisolone
- Rituximab + Chemotherapy (Active Comparator): In Part 2 only, participants will be randomized 1:1:1 to receive rituximab (R) with chemotherapy (CHOP), followed by rituximab monotherapy maintenance.
  Interventions: Drug: Odronextamab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prenisolone
- Odronextamab + Chemotherapy + Maintenance (Experimental): In Part 2, participants will be randomized 1:1:1 to receive odronextamab with chemotherapy [CHOP, or cyclophosphamide, vincristine, and prednisone (CVP)], followed by odronextamab monotherapy maintenance.
  Interventions: Drug: Odronextamab; Drug: Vincristine
- Odronextamab + Chemotherapy + No maintenance (Experimental): In Part 2, participants will be randomized 1:1:1 to receive odronextamab with chemotherapy (CHOP, or CVP) without maintenance.
  Interventions: Drug: Odronextamab; Drug: Vincristine

INTERVENTIONS:
Drug: Odronextamab — Administered by intravenous (IV) infusion
  Other Names: REGN1979
Drug: Rituximab — Administered by IV infusion, or subcutaneous (SC)
  Other Names: Rituxan
  Arms: Rituximab + Chemotherapy
Drug: Cyclophosphamide — Administered by IV infusion
  Other Names: Cytoxan
  Arms: Odronextamab + Chemotherapy; Rituximab + Chemotherapy
Drug: Doxorubicin — Administered by IV infusion
  Other Names: Adriamycin
  Arms: Odronextamab + Chemotherapy; Rituximab + Chemotherapy
Drug: Vincristine — Administered by IV infusion
  Other Names: Oncovin
  Arms: Odronextamab + Chemotherapy + Maintenance; Odronextamab + Chemotherapy + No maintenance; Rituximab + Chemotherapy
Drug: Prednisone/Prenisolone — Administered orally (PO)
  Other Names: Deltasone/Omnipred
  Arms: Odronextamab + Chemotherapy; Rituximab + Chemotherapy

SUMMARY:
This study is researching an experimental drug called odronextamab, referred to as study drug. The study is focused on participants with previously untreated follicular lymphoma. Follicular lymphoma is a type of non-Hodgkin lymphoma or NHL. Participants with follicular lymphoma that has come back after treatment (called "relapsed") or did not respond to treatment (called "refractory") are eligible to take part only in Part 1A of the study.

This study is made up of 3 parts: Part 1A (non-randomized), Part 1B and Part 2 (randomized - controlled).

The aim of Part 1A and Part 1B of the study is to see how safe and tolerable the study drug in combination with chemotherapy is and to determine the dose and schedule of the study drug to be combined with chemotherapy to be used in Part 2 of the study.

The aim of Part 2 of the study is to assess how effective the combination of the study drug with chemotherapy is in comparison with the combination of rituximab and chemotherapy (the current standard-of-care for NHL). Standard-of-care means the usual medication expected and used when receiving treatment for a condition.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)
* The impact from the study drug on quality-of-life and ability to complete routine daily activities

ELIGIBILITY:
Key Inclusion Criteria:

1. Have diagnosis of cluster of differentiation 20 positive (CD20+) FL grade 1-3a, stage II bulky or stage III / IV

   1. For Part 1A: previously untreated participants who have Follicular Lymphoma International Prognostic Index (FLIPI)-1 score of 3 to 5, or R/R FL
   2. For Part 1B: previously untreated participants who have FLIPI-1 score of 3 to 5
   3. For Part 2: previously untreated participants who have FLIPI-1 score of 0 to 5
2. Have measurable disease on cross sectional imaging documented by diagnostic computed tomography [CT], or magnetic resonance imaging [MRI] imaging, as described in the protocol
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
4. Adequate bone marrow and hepatic function.

Key Exclusion Criteria:

1. Participants with central nervous system lymphoma or leptomeningeal lymphoma
2. Participants with histological evidence of transformation to a high-grade or diffuse large B-cell lymphoma
3. Participants with Waldenström macroglobulinemia (WM, lymphoplasmacytic lymphoma), grade 3b follicular lymphoma, chronic lymphocytic leukemia or small lymphocytic lymphoma
4. Recent major surgery and history or organ transplantation
5. A malignancy other than NHL unless the participant is adequately and definitively treated and any other significant active disease or medical condition that could interfere with the conduct of the study or put the participant at significant risk, as described in the protocol.

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2029-07-29 (Estimated); Study Completion 2029-07-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) for odronextamab in combination with chemotherapy | Up to 35 days
  Part 1, DLT period
Incidence of treatment-emergent adverse events (TEAEs) of odronextamab in combination with chemotherapy | Up to 2 years
  Part 1, Treatment period
Severity of TEAEs of odronextamab in combination with chemotherapy | Up to 2 years
  Part 1, Treatment period
Complete Response rate at 30 months (CR30) assessed by independent central review (ICR) | Up to 30 months
  Part 2

SECONDARY OUTCOMES:
Odronextamab concentrations in serum when administered with chemotherapy | Up to 30 months
  Part 1, Maintenance period and Part 2, Induction period
Odronextamab concentrations in serum when administered as monotherapy | Up to 30 months
  Part 1 and Part 2, Maintenance period
Incidence of anti-odronextamab antibodies (ADAs) | Up to 30 months
  Part 1 and Part 2
Titers of ADAs to odronextamab | Up to 30 months
  Part 1 and Part 2
Incidence of neutralizing antibodies (NAb) to odronextamab | Up to 30 months
  Part 1 and Part 2
Best overall response (BOR) as assessed by the investigator | Up to 30 months
  Part 1, end of Induction period and end of Maintenance period
Progression free survival (PFS) as assessed by ICR | Up to 5 years
  Part 2
CR30 as assessed by local investigator | Up to 30 months
  Part 2
Change in patient reported physical functioning scale scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Cancer-30 (EORTC-QLQ-C30) | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a global health status (GHS)/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
PFS as assessed by local investigator | Up to 5 years
  Part 2
Event-free survival (EFS) as assessed by ICR | Up to 5 years
  Part 2
EFS as assessed by local investigator | Up to 5 years
  Part 2
Overall Survival (OS) | Up to 5 years
  Part 2
BOR as assessed by local investigator | Up to 30 months
  Part 2
BOR as assessed by ICR | Up to 30 months
  Part 2
Duration of response (DOR) assessed by ICR | Up to 5 years
  Part 2
DOR as assessed by local investigator | Up to 5 years
  Part 2
Time to next anti-lymphoma treatment (TTNT) | Up to 5 years
  Part 2
Incidence of TEAEs | Up to 2 years
  Part 2
Severity of TEAEs | Up to 2 years
  Part 2
Change in patient reported health related quality of life (HRQoL) as measured by EORTC-QLQ-C30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Change in cancer disease as measured by EORTC-QLQ-C30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Change in treatment related symptoms as measured by EORTC-QLQ-C30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Change in patient-reported lymphoma disease as measured by the Lymphoma Subscale of the Functional Assessment of Cancer Treatment-Lymphoma (FACT-LymS) | Up to 5 years
  Part 2 The FACT-Lym lymphoma subscale (LymS) includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Change in treatment-related symptoms as measured by the FACT-LymS | Up to 5 years
  Part 2 The FACT-LymS includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Change in patient-reported general health status per EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | Up to 5 years
  Part 2 The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Change in patient-reported treatment side effects burden per Functional Assessment of Cancer Therapy-General Global Population Item 5 (FACT-G GP5) | Up to 5 years
  Part 2 A single item GP5 of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).
Change in Patient Global Impression of Severity (PGIS) | Up to 5 years
  Part 2 The PGIS includes a single-item to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days. Patients will choose the response that best describes the severity of their overall cancer symptoms with options on a 5-point scale ranging from 1 (No symptoms) to 4 (Very Severe).
Change in Patient Global Impression of Change (PGIC) | Up to 5 years
  Part 2 The PGIC item includes a single-item to assess how a patient perceives their overall change in health status since the start of study treatment. Patients will choose from response options on a 7-point scale ranging from 1 (Much Better) to 7 (Much worse); 1- Much Better, 2-Moderately Better, 3-A Little Better, 4-About the Same, 5-A Little Worse, 6-Moderately Worse, 7-Much Worse.
Change in score of the FACT-G GP5 item in the patient population | Up to 5 years
  Part 2 A single item GP5 of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (145):
- United States (9):
  - Boca Raton Clinical Research (BRCR) Global, Plantation, Florida
  - Investigative Clinical Research of Indiana, Noblesville, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Center for Oncology and Blood Disorders, Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Prohealth Care Inc, Waukesha, Wisconsin
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
- Austria (7):
  - Karl Landsteiner University Hospital St. Poelten, Sankt Pölten, Lower Austria
  - Medical University of Graz, Graz, Styria
  - Landeskrankenhaus Hochsteiermark, Leoben, Styria
  - Innsbruck Medical University, Innsbruck, Tyrol
  - Kepler University Hospital, Linz, Upper Austria
  - Universitatsklinik fur Kinder und Jungendheilkunde, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (6):
  - Universitair Ziekenhuis (UZ) Gent/ Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Verenigde Ziekenhuizen van Waas en Durme, Sint-Niklaas, Oost-Vlaanderen
  - Algemeen Ziekenhuis St Jan Brugge Oostende Av, Bruges, West-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Regional de la Citadelle, Liège
- Brazil (22):
  - Hospital Santa Izabel - Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - Hospital Sao Rafael, Salvador, Estado de Bahia
  - Ensino e Terapia de Inovacao Clinica Amo (Etica), Salvador, Estado de Bahia
  - Hospital Sirio Libanes Brasilia, Brasília, Federal District
  - Instituto DOr de Pesquisa e Ensino Df Star, Brasília, Federal District
  - Instituto Mario Pena de Ensino Pesquisa e Inovacao, Belo Horizonte, Minas Gerais
  - Centro Oncologico do Triangulo (COT) - Uberlandia, Uberlândia, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra o Cancer, Natal, Rio Grande do Norte
  - Instituto Tacchini de Pesquisa em Saude, Bento Gonçalves, Rio Grande do Sul
  - Instituto do Cancer em Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Hematologia e Oncologia, Joinville, Santa Catarina
  - Animi Unidade de Tratamento Oncologico Ltda, Lages, Santa Catarina
  - Fundacao Pio XII Hospital de Amor, Barretos, São Paulo
  - Amaral Carvalho Hospital, Jaú, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto, São Paulo
  - Instituto Nacional de Cancer Jose Alencar Gomes da Silva, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - AC Camargo Cancer Center, São Paulo
  - Clinical Hospital of Medicine School at Sao Paulo University, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo
- Chile (4):
  - Hospital Clinico Universidad de Los Andes, Santiago, Las Condes
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Centro Oncologia de Precision Universidad Mayor, Santiago, Santiago Metropolitan
  - Inmunocel, Santiago, Santiago Metropolitan
- Czechia (2):
  - University Hospital Hradec Kralove, Hradec Králové, North Central Czech Republic
  - University Hospital Brno, Brno, South Moravian
- France (14):
  - Cannes Hospital (Centre Hospitalier Cannes Simone Veil), Cannes, Alpes Maritimes
  - CHRU de Tours, Tours, Centre-Val de Loire
  - Institut de Cancerologie du Gard, Nîmes, Gard
  - Centre Hospitalier de Mont-de-Marsan, Mont-de-Marsan, Nouvelle-Aquitaine
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - The Novo Hospital North West Val Deoise, Cergy-Pontoise, Pontoise
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier de Lens (Centre Hospitalier Dr Schaffner dLens), Lens
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Sud - Hôpital Haut Lévêque, Pessac
  - CHU de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier de Saint Nazaire, Saint-Nazaire
  - Hopital Victor Dupouy Argenteuil, Argenteuil, Île-de-France Region
- Germany (2):
  - Stadtisches Krankenhaus Kiel, Kiel
  - MVZ fuer Haematologie und Onkologie Rhein-Kreis GmbH, Neuss
- Israel (7):
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
- Italy (15):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-Cesena
  - Azienda Ospedaliera Ordine Mauriziano Torino, Presidio Umberto I of Turin, Turin, Piedmont
  - Azienda Ospedaliera Universitario Policlinico Palermo, Palermo, Sicily
  - ASST Grande Ospedale Metropolitano Niguarda - Main Address, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Europeo di Oncologia, Milan
  - A.O.U. di Modena, Modena
  - Federico II University, Napoli
  - Azienda Ospedaliera di Perugia, Perugia
  - University of Pisa, Section of Hematology, Pisa
  - Azienda Ospedaliera Regionale San Carlo, Potenza
  - UO Ematologia Ravenna, Ravenna
  - Azienda Unita Sanitaria Locale Irccs Arcispedale Santa Maria Nuova, Reggio Emilia
  - Azienda Osperdaliero-Universitaria Policlinico Umberto 1, Rome
  - Azienda Sanitaria Universitaria del Friuli Centrale, Udine
- Poland (9):
  - Matopolskie Centrum Medyczne S.C., Krakow, Lesser Poland Voivodeship
  - Aidport, Skorzewo, Wielkopolska
  - Szpital Uniwersytecki Nr2 Bydgoszcz, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Building of the Non-Invasive Medicine Center, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. Mikolaja Kopernika w Lodzi (Copernicus Memorial Hospital), Lodz
  - Centrum Innowacyjnych Terapii Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy Warszawa, Warsaw
  - Szpital Szpecjalistyczny w Walbrzychu, Wałbrzych
- Spain (21):
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Parc Tauli Sabadell Hospital Universitari, Sabadell, Barcelona
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Cruces University Hospital (Hospital Universitario Cruces), Barakaldo, Bizkaia
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Quiron Salud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario Doctor Balmis Alicante, Alicante, Valencia
  - Hospital Universitario Lucus Augusti, Lugo
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Clinica Universidad de Navarra- Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University Multipal Wan Fang University, Taipei
- Thailand (2):
  - Chulalongkorn University, Bangkok, Krung Thep Maha Nakhon [Bangko]
  - Khon Kaen University, Khon Kaen
- Turkey (Türkiye) (12):
  - Ankara University Faculty of Medicine, Mamak, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Yenimahalle, Ankara
  - Gazi University, Ankara, Central Anatolia
  - VM Medical Park Mersin Hospital, Mezitli, Mersin
  - Sakarya University, Sakarya, Serdivan
  - Tekirdag Namik Kemal University Hospital, Tekirdağ, Suleymanpasa
  - Liv Hospital Ankara, Ankara
  - VKV American Hopital, Istanbul
  - Istanbul University, Istanbul
  - Erci̇yes Uni̇versi̇ty, Kayseri
  - Ondokuz Mayıs University, Samsun
  - Zonguldak Bulent Ecevit University, Zonguldak
- United Kingdom (4):
  - Royal Cornwall Hospital, Truro, Cornwall
  - The Hillingdon Hospitals NHS Foundation Trust, Uxbridge, London
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - NHS Grampian: Aberdeen Royal Infirmary, Aberdeen

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: OLYMPIA — https://olympiastudies.com/en-us